CLINICAL TRIAL: NCT04599309
Title: Real-time Detection of ctDNA and/or HPV DNA in High-risk Locally-advanced Head and Neck Squamous Cell Carcinoma (LA-HNSCC): The Pre-MERIDIAN (Molecular Residual Disease Interception in High-risk LA-HNSCC) Study.
Brief Title: Real-time Detection of ctDNA and/or HPV DNA in High-risk Locally-advanced Head and Neck Squamous Cell Carcinoma
Status: Active, not recruiting | Type: Observational
Sponsor: University Health Network, Toronto (Other)
Collaborators: Princess Margaret Hospital, Canada (Other)
Responsible Party: Sponsor
Other Study IDs: PRE-MERIDIAN; 20-5804 (Other: CAPCR ID)
Record Dates: First submitted 2020-10-18; First posted 2020-10-22 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-05

CONDITIONS: Cancer; Head and Neck Squamous Cell Carcinoma; Head and Neck Cancer
Keywords: Kinetics of ctDNA; Kinetics of HPV DNA; High-risk LA-HNSCC; Liquid Biopsy; Head and Neck; Molecular Profiling; Advanced Cancer
MeSH Terms: conditions — Neoplasms; Squamous Cell Carcinoma of Head and Neck; Head and Neck Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples collected serially for cfDNA and DNA extraction. Archived tumor sample collected for tumor genomic DNA analysis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- PRE-MERIDIAN: Patients with a histological or cytological diagnosis of LA-HNSCC of the oral cavity, oropharynx, hypopharynx, and larynx (stage III HPV positive or stage III-IV HPV negative). Patients who are candidates for standard definitive treatment such as surgery followed by radiotherapy +/- chemotherapy, or definite radiotherapy, or definite chemoradiotherapy.

SUMMARY:
This research study will include patients with high risk locally advanced head and neck squamous cell carcinoma (LA-HNSCC) of the oral cavity, oropharynx, hypopharynx or larynx and patients that are starting on standard definitive treatment. Patients with both stage III HPV positive and stage III HPV negative will be included. In this study, we aim to evaluate feasibility of ctDNA and/or HPV DNA detection in real time in high-risk LA-HNSCC.

DETAILED DESCRIPTION:
PRE-MERIDIAN aims to study the kinetics of ctDNA and HPV DNA after standard treatment in high-risk LA-HNSCC patients. This is an important study to understand their role in detecting MRD and determine optimal timing for ctDNA and HPV DNA quantification for future studies in immunotherapy.

We hypothesize that HPV DNA (in HPV+) +/- ctDNA detection in plasma after standard therapy may be quantified and monitored as MRD in high risk LA-HNSCC patients. We further hypothesize that detection of MRD in high risk LA-HNSCC after standard therapy may predict recurrence. Finally, we hypothesize that ctDNA time-to-clearance will be longer than 4-6 weeks after the end of treatment in some LA-HNSCC patients and therefore MRD may be further tested at 8-10 weeks after the end of standard therapy

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytological confirmed LA-HNSCC of the oral cavity, oropharynx, hypopharynx, or larynx.
* Stage III HPV Positive or Stage III-IV HPV negative.
* Availability of tumor sample
* Patients who are candidates for standard definitive treatment defined as:
* Surgery followed by radiotherapy +/- chemotherapy OR
* Definite radiotherapy OR
* Definite chemoradiotherapy.

Exclusion Criteria:

* Early stage HNSCC (I and II)
* Distant metastatic HNSCC

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with a diagnosis of high risk locally advanced head and neck squamous cell carcinoma (LA-HNSCC) of the oral cavity, oropharynx, hypopharynx or larynx and patients that are starting on standard definitive treatment.
Sampling Method: Non-Probability Sample
Enrollment: 35 (Actual)
Dates: Start 2020-10-15 (Actual); Primary Completion 2023-03-31 (Actual); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of high-risk LA-HNSCC patients with successful detection of ctDNA and/or HPV DNA in real time | Through study completion, up to 2 years
  ctDNA will be detected using Cancer Personalized Profiling by deep Sequencing (CAPP-Seq), a personalized bespoke NGS assay, or a similar approach. HPV DNA will be measured using digital PCR (dPCR) in all plasma samples from HPV+ LA-HNSCC patients included in this study.

SECONDARY OUTCOMES:
Correlation of presence of ctDNA +/- HPV DNA after standard treatment with shorter relapse-free survival (RFS), as assessed by comparison of baseline ctDNA +/- HPV DNA detection with time to relapse | Through study completion, up to 2 years
  ctDNA will be detected using Cancer Personalized Profiling by deep Sequencing (CAPP-Seq), a personalized bespoke NGS assay, or a similar approach. HPV DNA will be measured using digital PCR (dPCR) in all plasma samples from HPV+ LA-HNSCC patients included in this study.
Change in kinetics of ctDNA and/or HPV DNA over time after the end of standard definitive treatment and at recurrence, as assessed by ctDNA/HPV DNA analysis at sequential time points. | Through study completion, up to 2 years
  To provide preliminary data on the role of ctDNA and HPV DNA on detecting MRD in high-risk LA-HNSCC patients after standard treatment.
Selection of the best time-point to detect MRD after standard definitive therapy in HNSCC, as assessed by comparison of quantified ctDNA +/- HPV DNA at 4-6 weeks vs 8-10 weeks. | Through study completion, up to 2 years
  To provide preliminary data on the role of ctDNA and HPV DNA on detecting MRD in high-risk LA-HNSCC patients after standard treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Lillian Siu, Principal Investigator — Princess Margaret Cancer Centre; Scott Bratman, Principal Investigator — Princess Margaret Cancer Centre
Locations (1):
- Princess Margaret Cancer Centre, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided
Targeted gene sequencing results, along with limited clinical information that does not identify the patient as an individual, such as age, partial date of birth (year, month), gender, cancer type, and pathology information related to the samples tested, and survival time may be shared with collaborating researchers.
  Data from this study can be shared through two types of databases: open-access or controlled-access. An open-access database is publicly accessible and contains limited clinical information and analyses of samples. A controlled-access database contains more detailed clinical information, such as relevant past medical history and the results of prior and ongoing cancer treatments, and analyses of samples, but is only accessible to researchers who sign agreements defining how data may be used. All data will be stripped of all personal identifying information.